CLINICAL TRIAL: NCT07279311
Title: Virtual Reality-enhanced Psychotherapy as a Mental Health Intervention During Antepartum Hospitalization: A Pilot Randomized Controlled Trial
Brief Title: Virtual Reality-enhanced Psychotherapy for Perinatal Depression
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Danielle Panelli, Instructor in Obstetrics & Gynecology - Maternal Fetal Medicine, Principal Investigator, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 79808
Record Dates: First submitted 2025-12-01; First posted 2025-12-12 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Depression During Pregnancy
Keywords: pregnancy; high risk pregnancy; antepartum hospitalization; depression; maternal mental health; virtual reality
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of care (No Intervention): Participants will receive standard therapy during their antepartum hospitalization, which will include consultations with social workers and psychiatry physicians (if recommended by the social worker).
- Virtual-Reality Behavioral Activation (Experimental): Participants will receive the 3-week VR-BA psychotherapy. The VR-BA consists of 4 self-guided VR sessions per week and a weekly telemedicine guided BA session with a trained study team member via ZOOM (and Spanish interpreter, if required) lasting 30-50 minutes. This will be a total of 3 telemedicine-guided BA sessions and 12 self-guided VR sessions over the course of the study.
  Interventions: Behavioral: Virtual reality behavioral activation

INTERVENTIONS:
Behavioral: Virtual reality behavioral activation — The available VR-BA sessions include immersive 360° videos using headsets. The content encompasses a wide range of categories, including but not limited to animals; sports, dance, or arts; adrenaline; travel; and hiking or the outdoors. The patient will select activities which align most with their values and interests, with guidance during the telehealth sessions. The videos range from 1 minute to 10 minutes.
  Arms: Virtual-Reality Behavioral Activation

SUMMARY:
Perinatal depression is a growing public health crisis in the United States, affecting one in five individuals during pregnancy or postpartum. Mental health conditions contribute to 23% of maternal deaths, underscoring the urgent need for innovative interventions. Obstetric patients who experience complications requiring prolonged hospitalization are particularly vulnerable to mental health deterioration. Virtual reality (VR) has shown promise for expanding access, reducing barriers, and enhancing first-line depression treatment when paired with evidence-based psychotherapies such as behavioral activation (BA). However, traditional BA is not feasible for inpatients, as their hospitalization prevents participation in conventional in-person, mood-boosting activities; VR-enhanced BA (VR-BA) presents a novel opportunity to address this gap.

The goal of the study is to compare a 3-week VR-BA protocol to standard therapy (social work consultation) for hospitalized pregnant individuals with depressive symptoms. The objectives are to assess 1) whether VR-BA is acceptable, tolerable, and feasible in this population and 2) whether it leads to greater reductions in depressive symptoms compared to standard therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to Stanford Children's Hospital antepartum unit for obstetric indications that are likely to warrant >3 weeks of hospitalization (such as vasa previa, preterm premature rupture of membranes, severe preeclampsia).
* Able to read and write in English or Spanish
* Baseline EPDS score on admission >=10 on routine screening
* Admitted >24 hours prior to enrollment

Exclusion Criteria:

* Patients with serious neuropsychiatric illness (bipolar disorder, schizophrenia, epilepsy, or suicidal ideation)
* Known delivery planned within the next 3 weeks

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-09 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Depressive symptoms scale score using Edinburgh Postnatal Depression Scale (EPDS) | At enrollment, then weekly up to a total of 3 weeks
  Edinburgh Postnatal Depression Scale (EPDS) scores will be compared at the end of the 3 week intervention between groups. The EPDS is a 10-item questionnaire, with total score 0-30. Higher scores are consistent with greater levels of depressive symptoms.

SECONDARY OUTCOMES:
Feasibility - dropout rate | Weekly, up to 3 weeks
  Number of participants who withdraw from the study (after enrollment) divided by total enrollment number
Feasibility - compliance rate | Weekly, up to 3 weeks
  Percentage of patients who complete VR-BA 4 sessions per week (total of 12).
Feasibility - adverse event rate | 3 weeks
  Occurrence of any of the following during the study: nausea, falls, seizure, suicidal ideation.
Acceptability - Presence Questionnaire | Weekly, up to 3 weeks
  Validated questionnaire (3 questions) asking about perception of the virtual reality experience using the headset and videos. Each response is rated on a Likert scale ranging from 0-4, with 0 being "not at all" and 4 being "very strongly".
Acceptability - Technology Acceptance Model | Weekly, up to 3 weeks
  Validated questionnaire (13 questions) asking participants about perceived usefulness, perceived ease of use, attitudes toward use, intention to use technology. Each response is rated on a Likert scale ranging from 0-4, with 0 being "strongly disagree" and 4 being "strongly agree".
Tolerability - Simulator Sickness Questionnaire | Weekly, up to 3 weeks
  Validated questionnaire (16 questions) asking participants about tolerability of wearing the headset. Each response is rated on a Likert scale ranging from 0-3, with 0 representing "no more than usual" and 3 representing "severely more than usual".

CONTACTS AND LOCATIONS:
Overall Officials: Danielle M Panelli, MD MS, Principal Investigator — Stanford University
Locations (1):
- Lucile Packard Children's Hospital, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No